CLINICAL TRIAL: NCT00950001
Title: Efficacy of Post-Surgical Stereotactic Radiosurgery for Metastatic Brain Disease: A Randomized Trial
Brief Title: Stereotactic Radiosurgery Compared to Observation in Treating Patients With Brain Metastases
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0381; NCI-2011-00542 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2009-0381 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (SRS) (Experimental): Patients undergo stereotactic radiosurgery to the surgical cavity within 30 days of the craniotomy.
  Interventions: Radiation: Stereotactic Radiosurgery
- Arm II (observation) (No Intervention): Patients undergo clinical observation after craniotomy.

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; stereotactic radiation therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
  Arms: Arm I (SRS)

SUMMARY:
This randomized phase III trial studies stereotactic radiosurgery to see how well it works compared to clinical observation after surgery in treating patients with brain metastases. Stereotactic radiosurgery, a type of radiation therapy, may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate benefit of post-surgical stereotactic radiosurgery (SRS) on the resection bed in providing 6 month local control (decreasing the risk of local tumor recurrence) when compared to surgical resection alone.

SECONDARY OBJECTIVES:

I. Overall survival, development of distant brain metastases and complications related to treatment.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo stereotactic radiosurgery to the surgical cavity within 30 days of the craniotomy.

ARM II: Patients undergo clinical observation after craniotomy.

After completion of study treatment, patients are followed up at 5-8 weeks, every 6-9 weeks for 1 year, every 3-4 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be older than 3 years of age (radiosurgical frames cannot be placed on children younger than age 3).
2. Patients must have 3 or fewer newly diagnosed metastatic lesions in the brain with a complete resection of at least one lesion as determined the study neuroradiologist.
3. The resection cavity must have a maximum diameter of less than or equal to 4cm. This criteria will be determined by the study radiologist.
4. Additional unresected brain metastases (up to 2) must have a maximum diameter of less than or equal to 3 cm.
5. Patients must be considered candidates for SRS within 30 days of surgical resection.
6. Patients must have a Karnofsky Performance Scores (KPS) of at least 70 at the first post operative visit. Patients under 18 years of age must have a Lansky Performance Score of of at least 70.
7. Patients must be able to undergo an MRI scan.
8. Patients must agree to randomization as documented by signing the Institutional Review Board (IRB) approved consent form.

Exclusion Criteria:

1. Patients who have received prior radiation therapy to the brain for any reason.
2. There is radiographic evidence of leptomeningeal disease prior to study entry.
3. The primary tumor is small-cell lung cancer, lymphoma, leukemia, or multiple myeloma.
4. For females, if they are pregnant or breast-feeding (The exclusion is made because gadolinium may be teratogenic in pregnancy).

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2009-08-13 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Time to local recurrence | 6 months
  A univariate test between groups will be conducted using a log rank test of Kaplan-Meier survival estimates and multivariate analyses will be conducted via the Cox proportional hazards model. The hazard ratio comparing each arm will be computed for each endpoint with and without adjustment for other covariates. Confidence intervals (95%) will be computed for the hazard ratio estimates. The proportion of patients experiencing neurological complications will be computed via univariate and multivariate logistic regression analysis.

SECONDARY OUTCOMES:
Overall survival | Up to 8 years
  A univariate test between groups will be conducted using a log rank test of Kaplan-Meier survival estimates and multivariate analyses will be conducted via the Cox proportional hazards model. The hazard ratio comparing each arm will be computed for each endpoint with and without adjustment for other covariates. Confidence intervals (95%) will be computed for the hazard ratio estimates.
Development of distant brain metastases | Up to 8 years
  A univariate test between groups will be conducted using a log rank test of Kaplan-Meier survival estimates and multivariate analyses will be conducted via the Cox proportional hazards model. The hazard ratio comparing each arm will be computed for each endpoint with and without adjustment for other covariates. Confidence intervals (95%) will be computed for the hazard ratio estimates.
Incidence of complications related to treatment | Up to 8 years
  The proportions of patients experiencing neurological complications will be computed via univariate and multivariate logistic regression analysis. The proportion of complications resulting in prolongation of hospital stay will also be computed. The odds ratios comparing both arms will be computed with and without adjustment for other covariates. Confidence intervals (95%) will be computed for the odds ratio estimates.
Proportion of patients experiencing neurological complications | Up to 8 years
  Computed via univariate and multivariate logistic regression analysis.
Proportion of complications resulting in prolongation of hospital stay | Up to 8 years
  Will be computed.
Time to first neurological complication | Up to 8 years
  A univariate test between groups will be conducted using a log rank test of Kaplan-Meier survival estimates and multivariate analyses will be conducted via the Cox proportional hazards model. The hazard ratio comparing each arm will be computed for each endpoint with and without adjustment for other covariates. Confidence intervals (95%) will be computed for the hazard ratio estimates.

CONTACTS AND LOCATIONS:
Overall Officials: Debra NAna Yeboa, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Mahajan A, Ahmed S, McAleer MF, Weinberg JS, Li J, Brown P, Settle S, Prabhu SS, Lang FF, Levine N, McGovern S, Sulman E, McCutcheon IE, Azeem S, Cahill D, Tatsui C, Heimberger AB, Ferguson S, Ghia A, Demonte F, Raza S, Guha-Thakurta N, Yang J, Sawaya R, Hess KR, Rao G. Post-operative stereotactic radiosurgery versus observation for completely resected brain metastases: a single-centre, randomised, controlled, phase 3 trial. Lancet Oncol. 2017 Aug;18(8):1040-1048. doi: 10.1016/S1470-2045(17)30414-X. Epub 2017 Jul 4. PMID 28687375
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org